CLINICAL TRIAL: NCT03836027
Title: Fertility Preservation and Reproductive Needs of Transgender People: Desires, Attitude and Knowledge of Subjects With Gender Dysphoria
Brief Title: Fertility Desires and Reproductive Needs of Transgender People
Acronym: PaFer
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03374-51
Record Dates: First submitted 2019-01-28; First posted 2019-02-11 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2020-07

CONDITIONS: Fertility Preservation; Parenting; Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Majority of transgender and gender nonconforming people seeking medical care are in pubertal and reproductive age. Cross-sex hormones may compromise fertility especially when preceded by puberty blocking regimen. Our current understanding on reproductive needs of transgender persons is insufficient.

The guidelines of Endocrine Society and the World Professional Association for Transgender Health prompt the health professionals to provide information on fertility risk and fertility preservation options before initiating hormonal treatment. Currently, no clear tools are available for healthcare professionals. Among several challenges for clinical care are a low clinical awareness, a lack of suitable psycho-educational instruments addressing fertility values that can be used to facilitate discussion between transgender persons and healthcare providers, a lack of established methods for fertility preservation in prepubertal youth, and a lack of long-term data regarding reproductive function, psychological and societal outcomes in this population. Likewise, current data are sparse regarding the experience of transgender and gender nonconforming people with fertility preservation.

Our aim is to describe desires, attitudes and knowledge of transgender and gender nonconforming people regarding fertility preservation wishes and reproductive needs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Follow-up in the Department of Endocrinology, Diabetology and Nutrition of the University Hospital of Nancy
* Gender dysphoria according to the ICD 11
* Voluntary, informed consent to participate in research
* Compulsory affiliation to the social security system

Exclusion Criteria:

-Refusal or incapacity to be involved in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participation to the study will be proposed consecutively to all subjects, fulfilling inclusion criteria, attending in-office follow-up visit for gender dysphoria in the Department of Endocrinology, Diabetology and Nutrition of the University Hospital of Nancy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Reproductive desires and attitudes of transgender and gender nonconforming people towards fertility preservation | 1 year
  A cross-sectional anonymous survey developed in the University Hospital of Nancy. Content validity of the questionnaire is endorsed by 2 endocrinologists specialized in transgender health (EF, VP). The first part provides general information on the characteristics of respondents (9 items). The second part concerns knowledge on fertility preservation (10 items), parental desires and constraints (8 items) and attitudes on fertility preservation issues (6 items). A descriptive analysis of the sample will be done using mean and standard deviation (or median and interquartile range) for quantitative variables, and counts and percentages for qualitative variables. The approval by the Institutional Review Board of the University Hospital of Nancy and the registration at French National Commission for Data Protection and Liberties are underway.

SECONDARY OUTCOMES:
Knowledge of subjects with gender dysphoria on the options of fertility preservation | 1 year
  Description of the construct and its evaluation is detailed in the section "primary outcome measure" as follows:
  A cross-sectional anonymous survey developed in the University Hospital of Nancy. Content validity of the questionnaire is endorsed by 2 endocrinologists specialized in transgender health (EF, VP). The first part provides general information on the characteristics of respondents (9 items). The second part concerns knowledge on fertility preservation (10 items), parental desires and constraints (8 items) and attitudes on fertility preservation issues (6 items). A descriptive analysis of the sample will be done using mean and standard deviation (or median and interquartile range) for quantitative variables, and counts and percentages for qualitative variables. The approval by the Institutional Review Board of the University Hospital of Nancy and the registration at French National Commission for Data Protection and Liberties are underway.
generic quality of life: physical functioning, limitations due to physical state, pain, mental health, limitations due to mental state, social health, vitality and global health | 1 year
  Questionnaire (Short form 36 health survey) The SF-36 is a generic quality of life self-questionnaire with 36 items grouped in 8 dimensions (physical functioning, limitations due to physical state, pain, mental health, limitations due to mental state, social health, vitality and global health). For each dimension a quality of life score is calculated and normalized between 0 (worst possible QoL) and 100 (best QoL possible).
Anxiety: State-Trait Anxiety Inventory, STAI-Y | 1 year
  * The STAI-Y assesses anxiety as a personality trait and as a specific emotional response to a situation. The first part, STAI-Y-1, consists of 20 sentences assessing the current emotional state of the subject. The second part, STAI-Y-2, consists of 20 sentences assessing the subject's usual emotional state.
  * Each answer to an item in the STAI-Y is scored from 1 to 4, with 1 indicating the lowest degree of anxiety and 4 the highest degree of anxiety.
  * In the STAI-Y-1, the subject indicates the intensity of his feelings on a 4-point Likert scale ranging from "not at all" to "many". In the STAI-Y-2, the subject indicates on a 4-point Likert scale ranging from "almost never" to "almost always", a frequency at which he usually feels the symptoms listed.
  * To obtain the score for the STAI-Y-1, the scores for the 20 items (1 to 20) are summed. To obtain the STAI-Y-2 score, the scores for the 20 items (21 to 40) are summed. Each score can therefore vary from 20 to 80.
Self-esteem : Physical self inventory, 25 items (PSI-25) | 1 year
  * The PSI-25 is an inventory of self-esteem relating to the body domain.
  * This tool consists of 6 scales: at the general level, the overall self-esteem scale, at the physical domain level: the perceived physical value scale, and at the subdomain level, 4 subscales: the fitness, athletic competence, physical appearance and strength. It has 25 items
  * The subject responds on the Likert scale in 6 increasing degrees (it looks like me 1: not at all, 2: very little, 3: a little, 4: enough, 5: a lot, 6: quite).
  * The score ranges from 5 to 30 for each scale, total score is averaged.
Depression: Center for Epidemiologic Studies Depression Scale, CES-D | 1 year
  * The CES-D assesses the frequency and severity of depressive symptoms presented by the general population. The questionnaire has 20 items.
  * The subject indicates on a 4-point Likert scale ranging from "almost never" to "almost always", a frequency at which he usually feels the symptoms listed.
  * Score is calculated from 0 to 60 (maximum score indicating strong expression of symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes